CLINICAL TRIAL: NCT01019967
Title: A Magnetic Resonance Spectroscopic Examination of Children and Adolescents Taking Riluzole for Obsessive-Compulsive Disorder
Status: Terminated | Type: Observational
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 100024; 10-M-0024
Record Dates: First submitted 2009-11-24; First posted 2009-11-25 (Estimated); Last update posted 2017-10-06 (Actual); Status verified 2012-09-20

CONDITIONS: Childhood Obsessive-Compulsive Disorder; Autism Spectrum Disorders
Keywords: Children and Adolescents; Obsessive-Compulsive Disorder; Magnetic Resonance Spectroscopy; Autism; OCD; Obsessive Compulsive Disorder
MeSH Terms: conditions — Autism Spectrum Disorder; Obsessive-Compulsive Disorder; Autistic Disorder

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Background:

* Obsessive-compulsive disorder (OCD) is a common childhood disorder that often does not respond to standard treatments. Researchers are exploring the role that a brain chemical called glutamate plays in symptoms of OCD, and are testing a drug called riluzole that reduces glutamate to see if changing the levels of glutamate in the brain will help treat the disorder.
* Researchers are interested in using magnetic resonance spectroscopy (MRS), a type of magnetic imaging, to take pictures of various chemicals in the brain. MRS images will be used to detect changes in brain levels of glutamate in children taking riluzole.

Objectives:

- To use magnetic resonance spectroscopy to study the levels of glutamate in the brains of children and adolescents who have been taking riluzole.

Eligibility:

- Children and adolescents ages 7 to 17 who are enrolled in the current NIMH riluzole trial protocol (05-M-0225), who are able to lie still in the scanner for about an hour each time, and who are willing to have up to three MRS scans.

Design:

* Researchers will study some children/adolescents before they begin to take the study medication riluzole or placebo these children will have an MRS scan before starting the study medication. The scan will take about an hour.
* About 2 weeks after reaching the full dose on the study medication, participants will have a second hour-long MRS scan. Participants will have a third MRS scan after being on the study medication for 12 weeks.
* Some children who have already completed 12 weeks on riluzole or placebo, and are now taking riluzole, will have only one MRS scan.

DETAILED DESCRIPTION:
Objective

This study uses magnetic resonance spectroscopy (MRS) to measure the neurotransmitter glutamate in the anterior cingulate cortex (and, if tolerated, the left caudate nucleus and possibly the thalamus) in children and adolescents.

Study Population

All of the subjects will be participants in an ongoing double-blind placebo-controlled trial (05-M-0225) of a glutamate antagonist, the drug riluzole, for Obsessive-Compulsive Disorder (OCD). The subjects are male and female children and adolescents, ages 7-17 years. They will all have met criteria for clinically significant OCD and will have failed to benefit from standard-of-care treatments or have been unable to tolerate the treatments. Some of the subjects will also have a diagnosis on the autism spectrum.

Design

In one group of sixteen young people, glutamate will be measured in the anterior cingulate cortex at three points in time:

* at baseline, before starting riluzole or placebo;
* within ten to fourteen days of the baseline evaluation, after reaching full dose of the study drug (active drug or placebo) to which the sixteen subjects have just been randomized;
* at the end of the twelve weeks of the double-blind phase of the study.

In a second group of sixteen young people, all of whom are subjects in the open-label phase of the same study, glutamate will be measured (first) in the anterior cingulate cortex at a single point in time when each subject has achieved steady state on the open-label drug riluzole. If the subject tolerates additional time in the scanner, glutamate will also be measured in the left caudate and possibly in the left thalamus. Glutamate levels in this group will be correlated with change in OCD measures.

Outcome Measures

* In the first group, change in glutamate activity in anterior cingulate associated with active drug (riluzole) administration, as compared with change in glutamate activity for the subjects taking placebo.
* In the second group, correlation between serum riluzole level, glutamate activity (or flux) in anterior cingulate (and possibly in the caudate and thalamus), and therapeutic effect.

ELIGIBILITY:
* INCLUSION CRITERIA:

Subjects may be included in the study only if they meet all of the following criteria:

1. Male or female subjects, 7 to 17 years of age.
2. Female subjects of childbearing potential must be using a medically accepted means of contraception or must remain abstinent.
3. Each legal guardian must have a level of understanding sufficient to agree to all required tests and examinations. Each legal guardian must understand the nature of the study. Each legal guardian must consent to study protocol.
4. Subjects must fulfill DSM-IV criteria for (OCD) and have a CY-BOCS score of greater than 20. In the double-blind phase, subjects enrolled in the combined OCD and ASD cohort must also meet DSM-IV criteria for Pervasive Developmental Disorder as well as OCD.
5. Each subject already taking medicine must be taking usually effective doses of a medicine demonstrated to be effective in childhood OCD, must have been stable on that dose for at least six weeks, and must have no newly recognized or intolerable adverse effects from that medicine. Subjects who are currently not taking such a medication must have had adequate trial in the past of at least one medicine that has been shown to be effective for the symptoms of childhood OCD, and must have failed to see improvement or must have had intolerable adverse effects from the medicine.
6. Subjects must be able to swallow capsules.
7. Subject in this protocol will all be enrolled in the riluzole for childhood OCD protocol (NIH 05-M-0225).

EXCLUSION CRITERIA:

Subjects will be excluded from the study for any of the following reasons:

1. Presence of psychotic symptoms or lifetime history of schizophrenia, bipolar disorder, other psychotic disorder, or other serious unstable psychiatric illness. Medicially unstable due to binging, purging, or starvation.
2. Judged clinically to be at risk for suicide (suicidal ideation, severe depression, or other factors). Diagnosis of DSM-IV Major Depressive Disorder is not necessarily an exclusion criterion.
3. Disabling Tic Disorder requiring contraindicated medicines.
4. Female subjects who are pregnant, nursing, or unwilling to use effective contraception.
5. Serious unstable illnesses, including gastroenterologic, respiratory, cardiovascular (including ischemic heart disease), endocrinologic, neurologic, immunologic, or hematologic disease.
6. Renal or hepatic dysfunction that would interfere with excretion or metabolism of riluzole as evidenced by increase above upper limits of normal for BUN/creatinine, or more than two-fold elevation above upper limits of normal of serum transaminases (ALT/SGPT, AST/SGOT), gamma glutamate (GGT), or bilirubin.
7. Documented history of hypersensitivity or intolerance to riluzole.
8. DSM-IV Substance Abuse Disorder within the past 90 days or Substance Dependence Disorder within the past 5 years, or any use of tobacco.
9. Taking contraindicated drugs.
10. Unable to swallow capsules.
11. In addition, patients will not receive cognitive-behavior therapy during the period of the study.

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 17 (Actual)
Dates: Start 2009-11-17; Study Completion 2012-09-20

PRIMARY OUTCOMES:
Change in brain glutamate after adding riluzole vs. placebo

SECONDARY OUTCOMES:
Correlation between brain glutamate activity and riluzole level

CONTACTS AND LOCATIONS:
Overall Officials: Susan E Swedo, M.D., Principal Investigator — National Institute of Mental Health (NIMH)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Ajroud-Driss S, Saeed M, Khan H, Siddique N, Hung WY, Sufit R, Heller S, Armstrong J, Casey P, Siddique T, Lukas TJ. Riluzole metabolism and CYP1A1/2 polymorphisms in patients with ALS. Amyotroph Lateral Scler. 2007 Oct;8(5):305-9. doi: 10.1080/17482960701500650. PMID 17852022
- [Background] Arnold PD, Macmaster FP, Richter MA, Hanna GL, Sicard T, Burroughs E, Mirza Y, Easter PC, Rose M, Kennedy JL, Rosenberg DR. Glutamate receptor gene (GRIN2B) associated with reduced anterior cingulate glutamatergic concentration in pediatric obsessive-compulsive disorder. Psychiatry Res. 2009 May 15;172(2):136-9. doi: 10.1016/j.pscychresns.2009.02.005. Epub 2009 Mar 25. PMID 19324536
- [Background] Becquet D, Faudon M, Hery F. In vivo evidence for an inhibitory glutamatergic control of serotonin release in the cat caudate nucleus: involvement of GABA neurons. Brain Res. 1990 Jun 11;519(1-2):82-8. doi: 10.1016/0006-8993(90)90063-h. PMID 1975768